CLINICAL TRIAL: NCT05148767
Title: Neoadjuvant Chemoradiation With Irinotecan Guided by UGT1A1 Status in Patients With Locally Advanced Rectal Cancer: A Real-Word Multi-center Study
Brief Title: UGT1A1-Based Irinotecan Therapy for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, MD, Chief physician, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG-2003
Record Dates: First submitted 2021-10-07; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Rectal Cancer Stage III
Keywords: locally advanced rectal cancer; Neoadjuvant chemoradiotherapy; irinotecan
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant chemoradiotherapy based on irinotecan (Experimental): Locally advanced rectal cancer patients who were treated with irinotecan-based neoadjuvant chemoradiotherapy regimen can be enrolled in this group.
  Interventions: Drug: Neoadjuvant chemoradiotherapy based on irinotecan

INTERVENTIONS:
Drug: Neoadjuvant chemoradiotherapy based on irinotecan — Patients with locally advanced rectal cancer treated with irinotecan-based chemoradiotherapy were enrolled in this study. The dose of irinotecan is determined by the genotype of UGT1A1.Concurrent Chemoradiotherapy:
  Radiation: 50Gy/25Fx; Capecitabine: 625mg/m2 bid Monday-Friday per week; Irinotecan: 80mg/m2 (UGT1A1*28 and *6: 6/6+GG) or 65mg/m2 (UGT1A1*28 and *6 ：6/7+GG or 6/6+GA) or 50mg/m2 （UGT1A1*28 and *6 ：7/7+GG or 6/6+AA or 6/7+GA）.

SUMMARY:
To explore whether the application of irinotecan under the guidance of UGT1A1 gene in neoadjuvant chemotherapy and radiotherapy for locally advanced rectal cancer could improve the clinical efficacy in the real world.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiotherapy (nCRT) combined with surgery is the standard care of treatment for locally advanced rectal cancer (LARC), which could effectively reduce the risk of local recurrence, increase the chance of sphincter preservation, and effectively improve the quality of life of patients. However, only about 8% of patients can benefit from nCRT. Therefore, to improve the therapeutic effect of nCRT and retain the organ function of patients so as to improve their quality of life is the focus of the current investigation.

In the previous study, the investigator have completed a series of clinical researches of irinotecan guided by UGT1A1 gene for nCRT in rectal cancer. A dose climbing study was firstly conducted to explore the maximum tolerable dose of irinotecan for nCRT in rectal cancer. The results indicated that the weekly dose intensity of irinotecan could be increased from 50mg/m2 to 80mg/m2 when the genotype of UGT1A1*28 locus was 6/6, and the weekly dose intensity of irinotecan could also reach 65mg/m2 when the genotype of irinotecan was 6/7 phenotype. Further analysis also demonstrated that there was a dose-effect relationship between the total dose of irinotecan and pathological complete remission (pCR). The recently published CinClare study is a 3-phase randomized controlled trial that doubles the pCR rate and the total CR rate in combination with irinotecan on the basis of capecitabine combined with radiotherapy. However, in the Aristotle study conducted in the United Kingdom at the same phase, it has not been proved that irinotecan could improve the pCR rate, and it is not known whether the difference between the two studies is completely attributed to the irinotecan dose. Therefore, the investigator designed this real-world study to explore whether irinotecan can indeed improve the treatment efficacy in the real world when using irinotecan under the guidance of UGT1A1 gene in nCRT for LARC. Any locally advanced rectal cancer patients treated with irinotecan-based neoadjuvant radiotherapy and chemotherapy can be enrolled in this study. It is expected that the results of this study could provide more basis for individualized treatment of LARC.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed rectal adenocarcinoma
2. Clinical stage T3-4 and / or Nude positive, and the treatment plan is nCRT.
3. Without distance metastases
4. A need for tumor withdrawal.
5. Aged 18-75 years old, regardless of gender.
6. ECOG score 0-2.
7. Detection of UGT1A1*6 and * 28 gene status.
8. Be able to comply with the plan during the study period.
9. Sign the inform consent

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Those with other history of malignant disease in the past 5 years, except for cured skin cancer and cervical carcinoma in situ
3. If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
4. Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention (see appendix 12), or a history of myocardial infarction in the last 12 months
5. Organ transplantation requires immunosuppressive therapy Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
6. Subject blood routine and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; Alanine transaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal; alkaline phosphatase (ALP) ≤2.5 times the normal upper limit; serum total bilirubin <1.5 times the normal upper limit; serum creatinine <1 times the normal upper limit; serum albumin ≥ 30g / L
7. Anyone who is allergic to any research medication
8. DPD deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 3 months after neoadjuvant chemoradiotherapy
  The tumor disappeared completely and the tumor markers remained normal for at least 4 weeks.
Locally recurrence rate | Within 5 years after the end of treatment
  The proportion of recurrent rectal tumors in the total population after the complete regression of rectal tumors
DFS | Within 5 years after the end of treatment
  The time from complete regression of the tumor after neoadjuvant therapy or radical resection to the first recurrence or death
OS | Within 5 years after the end of treatment
  The time from enrolled in the study to death caused by any cause
Toxicity effect | Within 5 years after the end of treatment
  Any adverse reactions caused by neoadjuvant chemoradiotherapy or surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ji Zhu, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China